CLINICAL TRIAL: NCT06552845
Title: Exploratory Study of Consistency of Bi-Atrial Fibrosis Detected by Late Gadolinium Enhancement Magnetic Resonance Imaging and Low Voltage Area of Electroanatomic Mapping
Brief Title: Consistency of LGE-MRI Fibrosis and EAM Low-voltage Area
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-2223
Record Dates: First submitted 2024-08-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Inclusion Criteria
  1. Adult patients (≥18 years old) who are willing to participate in this study and can sign informed consent;
  2. Atrial fibrillation was diagnosed and catheter ablation was proposed Exclusion criteria
  a) Left atrial thrombus or left atrial appendage thrombus; b) Severe chronic obstructive pulmonary disease (FEV1/ FVC<70%, FEV1<50% predicted value); c) Absolute contraindications of anticoagulation therapy; d) Currently pregnant; e) Contraindications for LGE-MRI (claustrophobia, pacemaker implantation, eGFR<30ml/min for renal insufficiency, severe obesity, pregnancy, gadolinium chelating agent allergy, etc.); f) refuse to participate in the study; g) other physical or mental incapacity to participate in the study.
  Interventions: Diagnostic Test: LGE-MRI Scan

INTERVENTIONS:
Diagnostic Test: LGE-MRI Scan — Participants will receive LGE-MRI scan before catheter ablation and 3 months after catheter ablation

SUMMARY:
This study aims to:

1. Assess the consistency of LGE-MRI bi-atrial fibrosis and electroanatomical mapping of bi-atrial low voltage region
2. To evaluate the electroanatomical characteristics of different types of fibrosis (dense fibrosis, patchy fibrosis, etc.) in different locations of the left and right atrium;
3. To explore the correlation between preoperative and postoperative bi-atrial fibrosis and long-term recurrence in patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years old) who are willing to participate in this study and can sign informed consent;
2. Atrial fibrillation was diagnosed and catheter ablation was proposed

Exclusion Criteria:

1. Left atrial thrombus or left atrial appendage thrombus;
2. Severe chronic obstructive pulmonary disease (FEV1/ FVC<70%, FEV1<50% predicted value);
3. Absolute contraindications of anticoagulation therapy;
4. Currently pregnant;
5. Contraindications for LGE-MRI (claustrophobia, pacemaker implantation, eGFR<30ml/min for renal insufficiency, severe obesity, pregnancy, gadolinium chelating agent allergy, etc.);
6. refuse to participate in the study;
7. other physical or mental incapacity to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult AF patients who are planned to receive catheter ablation and have no contraindications of LGE-MRI
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Consistency of LGE-MRI fibrosis and EAM low-voltage area | Baseline (at recruit time point)
  Use Registration to match the corresponding spatial points of LGE-MRI and EAM。Each spatial points will contain two types of status(Fibrosis: Yes/No, Low-voltage area: Yes/No). Chi-square test will be used to assess the consistency of fibrosis and low-voltage area.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, CAMS&PUMC, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared under the permission of primary investigator